CLINICAL TRIAL: NCT05633914
Title: A Phase II Study of Tucidinostat and Nab-paclitaxel in Advanced HR+/HER2- Breast Cancer
Brief Title: Tucidinostat and Nab-paclitaxel in Advanced HR+/HER2- Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C34
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: HR+/HER2- Breast Cancer
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat and nab-paclitaxel (Experimental)
  Interventions: Drug: Tucidinostat; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Tucidinostat — 20mg, po., biw, q3w
  Other Names: Chidamide
Drug: nab-paclitaxel — 125mg/m2, d1, iv.drip, q7d
  Other Names: ABRAXANE

SUMMARY:
This study is looking to see whether the combination of Tucidinostat and nab-paclitaxel is safe and effective in participants with advanced HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, ≤75, female;
2. Histologically confirmed HR positive and HER2 negative postmenopausal metastatic breast cancer patients [HER2 negative is defined as immunohistochemistry(IHC) 0 or IHC 1+, and if the score of IHC is 2+, fluorescence in situ hybridization technology (FISH) test must be negative, HR positve is defined as ER or PR ≥1%];
3. Primary endocrine resistance or at least experienced one line of endocrine therapy for recurrent or metastatic disease;
4. No more than 1 prior line of chemothrapy for recurrent or metastatic disease;
5. Patients who have been exposed to taxanes in neoadjuvant or adjuvant setting will be allowed to enroll, if they have obtained benifits from neoadjuvant treatment or have progressed ≥ 12 months from completion of adjuvant treatment;
6. ECOG performance status ≤ 1;
7. At least one measurable disease based on RECIST v1.1
8. Adequate organ function;
9. Life expectancy is more than 3 months;
10. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Prior exposed to histone deacetylase inhibitors, or received taxanes for metastatic disease;
2. Known hypersensitivity to any formulation component of the study drug;
3. Received chemotherapy, targeted therapy, Chinese herbal medicine with anti-tumor indications, or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 4 weeks before enrollment, or still within 5 half-lives of such drugs;
4. Toxicities that did not recover to National Cancer Institute Common Adverse Event Terminology Version 5.0 (NCICTCAEv5.0) grade 0 or 1 toxicity from prior antineoplastic therapy prior to the first dose of study treatment(alopecia, grade 2 fatigue, grade 2 anemia, non-clinically critical and asymptomatic laboratory abnormalities can be enrolled);
5. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
6. Pregnant or lactating female.
7. Any other conditions deemed inappropriate by the investigator to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  ORR by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Time from treatment until disease progression or death
Disease Control Rate （DCR） | 2 years
  the total proportion of patients with complete response（CR）, partial response（PR）and Stable Disease（SD）
Disease Control Rate （DCR） | 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No